CLINICAL TRIAL: NCT05216458
Title: Using Personalized Letters and Emails to Increase Health Insurance Take-up and Improve Plan Choice Quality in California's ACA Marketplace
Brief Title: Using Personalized Letters and Emails to Increase Health Insurance Take-up and Improve Plan Choice Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Office of Evaluation Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Feher, Research Scientist, Office of Evaluation Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05272021
Record Dates: First submitted 2021-12-31; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Health Behavior
Keywords: Affordable Care Act; randomized controlled trial; nudge; American Rescue Plan
MeSH Terms: conditions — Health Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Households in the control group did not receive any messages during the intervention period from June 2021 to August 2021
  Interventions: Behavioral: Control group
- Generic Outreach (Experimental): Households in the generic outreach group were assigned to receive a letter and two email reminders in June 2021 and thereafter received the standard messages Covered California sends to prospective enrollees, which explain that nearly all Covered California members get subsidies to pay for health insurance and encourage them to explore their plan options using an online Shop & Compare tool.
  For the generic arm, the outreach materials described new financial assistance under the American Rescue Plan and noted the availability of plans as low as $1/month.
  Interventions: Behavioral: Emails and letter intervention
- Personalized Outreach (Experimental): Households in the personalized outreach group were assigned to receive a letter and two email reminders in June 2021 and thereafter received the standard messages Covered California sends to prospective enrollees.
  For the personalized arm, the outreach explicitly informed the household that they were eligible for a $1/month CSR Silver 94 plan and described the benefits this plan confers. The outreach materials for the personalized group were not only designed to increase enrollment, but also to simplify the search process by providing households with a clear recommendation to pick a CSR Silver plan; this included highlighting the low out-of-pocket costs these plans provide when accessing care, a screenshot of what the plan would look like when they entered the shopping portal and peer comparison language that noted 9 out of 10 consumers like them choose CSR Silver plans
  Interventions: Behavioral: Emails and letter intervention

INTERVENTIONS:
Behavioral: Emails and letter intervention — Emails and letters for households assigned to the treatment group
  Arms: Generic Outreach; Personalized Outreach
Behavioral: Control group — No outreach during the intervention period.
  Arms: Control

SUMMARY:
With the passage of the American Rescue Plan (ARP) in March 2021, more consumers than ever before are now eligible for $0 -- or $1 per member per month (PMPM) in Marketplaces that include abortion coverage -- health insurance coverage across the ACA Marketplaces. But many individuals may not be aware of the new subsidies, or of their eligibility for Cost-Sharing Reduction (CSR) Silver plans. This project's goal is to examine whether personalized letters and email reminders can increase health insurance enrollment, CSR Silver take-up and $1 PMPM coverage.

ELIGIBILITY:
Inclusion Criteria:

* Submitted a Covered California application for the 2021 coverage year and found eligible for a $1 PMPM Enhanced Silver 94 plan

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44000 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percent of households enrolled in an ACA plan | Three months
  Percent of households enrolled in an ACA plan based on Covered California administrative data
Percent of households who chose a CSR Silver plan | Three months
  Percent of households in a CSR Silver plan based on Covered California administrative data
Percent of households who enrolled in a $1/month net-of-subsidy premium plan | Three months
  Percent of households who enrolled in a $1/month net-of-subsidy premium plan based on Covered California administrative data

SECONDARY OUTCOMES:
Percent of households who logged into their online account | Three months
  Percent of households who logged into their online account based on Covered California administrative data

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feher, PhD, Study Director — Covered California
Locations (1):
- Covered California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are committed to sharing as much data as possible for replication, consistent with the privacy and security requirements of the state agency that govern the re-disclosure of the data.
Supporting Information: SAP
Time Frame: Data will be available with investigator support upon publication.
Access Criteria: Replication data can be accessed via request to the primary investigator upon publication.

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT05216458/SAP_000.pdf